CLINICAL TRIAL: NCT00396799
Title: An Open-Label, Single-Dose, Randomized-to-Sequence, 2-Period, Crossover, Pivotal Bioequivalence Study Between Bazedoxifene Acetate/Conjugated Estrogens (Premarin Current Process) and Bazedoxifene Acetate/Conjugated Estrogens (Premarin New Process) Tablets Administered to Healthy Postmenopausal Women
Brief Title: Bioequivalence Study Of Bazedoxifene/Conjugated Estrogen Tablets In Postmenopausal Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3115A1-114
Record Dates: First submitted 2006-11-07; First posted 2006-11-08 (Estimated); Last update posted 2007-03-13 (Estimated); Status verified 2007-03

CONDITIONS: Menopause
MeSH Terms: interventions — bazedoxifene; Estrogens, Conjugated (USP)

INTERVENTIONS:
Drug: bazedoxifene/conjugated estrogens

SUMMARY:
The primary objective is to evaluate the bioequivalence between bazedoxifene/conjugated estrogens tablets produced using the current manufacturing process to bazedoxifene/conjugated estrogens tablets produced using a new manufacturing process

ELIGIBILITY:
Inclusion Criteria

* Healthy, postmenopausal women aged 35 to 70 years and weighing at least 50 kg (approx. 110 lbs).
* At least 6 months of spontaneous amenorrhea (with follicle-stimulating hormone levels of 39 mIU/mL or greater).
* Nonsmoker or smoker of fewer than 10 cigarettes per day, with ability to abstain for 5 days.

Exclusion Criteria

* Women with amenorrhea starting after 54 years of age.
* A history or active presence of clinically important medical diseases.
* Use of oral estrogen-, progestin, androgen-, or SERM-containing drug products within 30 days before receiving study drug.

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2006-11; Study Completion 2006-11

PRIMARY OUTCOMES:
Pharmacokinetic measures of blood levels of endogenous estrogen hormones, conjugated estrogens and bazedoxifene.

SECONDARY OUTCOMES:
Safety will be evaluated from reported signs and symptoms, scheduled physical examinations, gynecologic examinations, vital sign measurements, 12-lead ECG and clinical laboratory test results.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Principal Investigator — Wyeth is now a wholly owned subsidiary of Pfizer